CLINICAL TRIAL: NCT06216275
Title: Enhancing Calm in Arab Elderly With Dementia: Integrating Snoezelen Methods With Aromatherapy and Personal Items to Reduce Agitation
Brief Title: Enhancing Calm in Arab Elderly With Dementia
Acronym: sn/dm
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mostafa Shaban (Other)
Responsible Party: Sponsor-Investigator, Mostafa Shaban, Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Snoezelen_Demntia
Record Dates: First submitted 2024-01-08; First posted 2024-01-22 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Dementia; Agitation in Dementia, Including Alzheimer's Disease
Keywords: Dementia Care; Agitation in Elderly; Arab Elderly Dementia; Snoezelen Therapy; Aromatherapy in Dementia; Multi-sensory Stimulation
MeSH Terms: conditions — Dementia; Aberrant Motor Behavior in Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants receiving the integrated approach of Snoezelen therapy, aromatherapy, and the use of personal items.
  Interventions: Behavioral: Integrated Snoezelen-Aromatherapy-Personal Item Therapy
- Control Arm (No Intervention): Participants receiving standard care practices for dementia and agitation without the integrated approach.

INTERVENTIONS:
Behavioral: Integrated Snoezelen-Aromatherapy-Personal Item Therapy — Intervention Description:
  This unique intervention combines three distinct therapeutic approaches specifically tailored for Arab elderly patients with dementia experiencing agitation.
  Snoezelen Therapy: Customized sessions in a Snoezelen environment - a specialized room designed to deliver controlled multi-sensory stimuli. This room features adaptable lighting, colors, sounds, and textures to provide a soothing and stimulating experience. Sessions are personalized based on each patient's response and preference, under the guidance of trained professionals.
  Aromatherapy: Carefully selected essential oils known for their calming properties are used in a culturally sensitive manner. These oils are diffused in the environment or used during individual sessions to provide a relaxing olfactory experience. The choice of oils and method of delivery are standardized
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of integrating Snoezelen methods with aromatherapy and personal items in reducing agitation in Arab elderly individuals with dementia. The main questions it aims to answer are:

Does the combination of Snoezelen methods, aromatherapy, and the use of personal items significantly reduce agitation in elderly Arab patients with dementia compared to standard care practices? How do patients and caregivers perceive the impact of this integrated approach on the overall well-being and quality of life of the patients?

Participants in this study will:

Engage in sessions utilizing Snoezelen methods, a multi-sensory environment designed to deliver stimuli to various senses.

Receive aromatherapy treatments with selected scents known for their calming properties.

Be provided with personal items that are familiar and meaningful to them, to create a sense of comfort and security.

DETAILED DESCRIPTION:
This clinical trial is centered on a novel approach to dementia care, specifically targeting the Arab elderly demographic. It uniquely combines three elements - Snoezelen therapy, aromatherapy, and the use of personal items - to address agitation, a common and challenging symptom in dementia patients.

Snoezelen Therapy Implementation:

Custom-designed Snoezelen rooms will be used, equipped with lights, colors, sounds, and textures to stimulate senses in a controlled manner.

Sessions will be tailored to individual patient needs and preferences, monitored by trained staff.

Aromatherapy Application:

Selection of aromas will be based on their known calming properties, with a focus on cultural relevance and acceptability in the Arab elderly population.

The method of delivery and duration of each aromatherapy session will be standardized to ensure consistency across the study.

Incorporation of Personal Items:

Patients will be encouraged to select personal items that hold significant emotional value or are tied to pleasant memories.

These items will be integrated into the therapy sessions to provide a sense of familiarity and emotional comfort.

Data Collection and Analysis:

Quantitative data on agitation levels will be gathered using established agitation scales, both pre- and post-intervention.

The study aims to provide a comprehensive evaluation of how this integrated approach can influence agitation in dementia, considering both statistical effectiveness and personal experiences. The outcome will contribute valuable insights into dementia care practices, particularly for the Arab elderly population, and may offer a template for culturally sensitive dementia care.

ELIGIBILITY:
For the study "Enhancing Calm in Arab Elderly with Dementia: Integrating Snoezelen Methods with Aromatherapy and Personal Items to Reduce Agitation", here are the suggested Inclusion and Exclusion Criteria:

Inclusion Criteria:

* Age: Participants must be 65 years to 90 years
* Diagnosis: Clinical diagnosis of dementia required.
* Ethnicity: Must be of Arab descent.
* Agitation Levels: Must show agitation signs based on a standardized scale.
* Cognitive Function: Adequate cognitive function for study participation, verified by standard assessment.

Exclusion Criteria:

* Severe Medical Conditions: Individuals with severe medical conditions that could affect study participation or health.
* Advanced Dementia: Patients with very advanced dementia stages, unable to engage in study activities.
* Allergies: Known allergies to aromatherapy products used in the study.
* Recent Medication Changes: Significant changes in dementia medication regimen before the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Agitation Levels | 4 weeks
  The primary outcome measure is the reduction in agitation levels among the Arab elderly with dementia participating in the study. This will be quantitatively assessed using a validated agitation scale, such as the Cohen-Mansfield Agitation Inventory (CMAI) or a similar tool appropriate for dementia patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt

REFERENCES:
- [Background] Smith BC, D'Amico M. Sensory-Based Interventions for Adults with Dementia and Alzheimer's Disease: A Scoping Review. Occup Ther Health Care. 2020 Jul;34(3):171-201. doi: 10.1080/07380577.2019.1608488. Epub 2019 May 8. PMID 31066598
- [Background] Hogg J, Cavet J, Lambe L, Smeddle M. The use of 'Snoezelen' as multisensory stimulation with people with intellectual disabilities: a review of the research. Res Dev Disabil. 2001 Sep-Oct;22(5):353-72. doi: 10.1016/s0891-4222(01)00077-4. PMID 11580163
- [Background] Burns I, Cox H, Plant H. Leisure or therapeutics? Snoezelen and the care of older persons with dementia. Int J Nurs Pract. 2000 Jun;6(3):118-26. doi: 10.1046/j.1440-172x.2000.00196.x. PMID 11249409
- [Background] Merrick J, Cahana C, Lotan M, Kandel I, Carmeli E. Snoezelen or controlled multisensory stimulation. Treatment aspects from Israel. ScientificWorldJournal. 2004 May 11;4:307-14. doi: 10.1100/tsw.2004.30. PMID 15167944
- [Background] Chitsey AM, Haight BK, Jones MM. Snoezelen: a multisensory environmental intervention. J Gerontol Nurs. 2002 Mar;28(3):41-9. doi: 10.3928/0098-9134-20020301-09. PMID 11913515
- [Background] Carvalho SC, Martins FS, Martins AN, Barbosa RC, Vicente SG. Effectiveness of Snoezelen in older adults with neurocognitive and other pathologies: A systematic review of the literature. J Neuropsychol. 2024 Jun;18(2):312-331. doi: 10.1111/jnp.12346. Epub 2023 Sep 21. PMID 37735859
- [Background] Seegers H, Serani I, Bogar M, Gei M, Baudet V, Witz L, Bouchard JP. [The Snoezelen approach in pain management in psychiatry]. Soins Psychiatr. 2019 Jan-Feb;40(320):35-40. doi: 10.1016/j.spsy.2018.11.008. French. PMID 30654878
- [Background] Chung JC, Lai CK, Chung PM, French HP. Snoezelen for dementia. Cochrane Database Syst Rev. 2002;2002(4):CD003152. doi: 10.1002/14651858.CD003152. PMID 12519587
- [Background] Sigal A, Sigal M. The Multisensory/Snoezelen Environment to Optimize the Dental Care Patient Experience. Dent Clin North Am. 2022 Apr;66(2):209-228. doi: 10.1016/j.cden.2021.12.001. PMID 35365274
- [Derived] Alruwaili AN, Alruwaili MM, Ramadan OME, Ali SI, Shaban M. Nursing strategies for enhancing calm in older Arabs with dementia: integrating Snoezelen methods, aromatherapy, and personal items to reduce agitation. Geriatr Nurs. 2024 Sep-Oct;59:379-391. doi: 10.1016/j.gerinurse.2024.07.017. Epub 2024 Aug 10. PMID 39128143